CLINICAL TRIAL: NCT04473664
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics, Safety and Tolerability of Quizartinib in Subjects With Moderate Impaired Hepatic Function as Defined by NCI-ODWG Criteria
Brief Title: A Study of Quizartinib Pharmacokinetics in Participants With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-U105
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-09

CONDITIONS: Hepatic Impairment; Moderate Impaired Hepatic Function
Keywords: Hepatic Impairment; Healthy Subjects; Drug-drug Interaction; Pharmacokinetics; Quizartinib
MeSH Terms: interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment as defined by NCI-ODWG criteria who received a single, oral dose of quizartinib 30 mg on Day 1.
  Interventions: Drug: Quizartinib
- Control Participants with Normal Hepatic Function (Experimental): Healthy participants with normal hepatic function matched as a group by sex, age (±10 years), and weight (±20%) who received a single, oral dose of quizartinib 30 mg on Day 1.
  Interventions: Drug: Quizartinib

INTERVENTIONS:
Drug: Quizartinib — Single oral dose, 30 mg tablet

SUMMARY:
Quizartinib is a novel oral Class III receptor tyrosine kinase (RTK) inhibitor exhibiting highly potent and selective but reversible inhibition of Feline McDonough sarcoma (FMS)-like tyrosine kinase 3 (FLT3). Quizartinib is currently being studied alone or in combination with other agents as a treatment for acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) in adult and pediatric populations.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the plasma pharmacokinetics (PK) of quizartinib and its pharmacologically active metabolite AC886 after a single oral dose of 30 mg in participants with moderate hepatic impairment (HI) (as defined by National Cancer Institute-Organ Dysfunction Working Group [NCI-ODWG] criteria) compared to the healthy control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years to 75 years of age (inclusive), with a body mass index (BMI) of 18 kg/m^2 to 36 kg/m^2 (inclusive)
* In females, documented surgical sterilization, postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum at Screening), or agreement to use an approved form of contraception
* In males, documented surgical sterilization, sexual abstinence, or agreement to use an approved form of contraception from Screening until 6 months after the dose of quizartinib
* In males, agreement to avoid sperm donation for 6 months days after the dose of quizartinib
* Participants must agree to refrain from donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, and platelets from 6 weeks prior to Screening.
* All participants must be willing to refrain from consuming grapefruit/grapefruit juice, Seville oranges, and pomegranates/pomegranate juice 10 days before the dose of the study drug is given on Day 1 until end-of-study.

Exclusion Criteria:

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormality) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures
* Laboratory results (serum chemistry, hematology, and urinalysis) outside the normal range, if considered clinically significant by the investigator Estimated glomerular filtration rate (eGFR) < 90 mL/min at screening.
* Women who are pregnant or breastfeeding
* Use of any drugs or substances known to be inhibitors or inducers of CYP3A4/5 within 28 days from the first dose or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to quizartinib administration and during the study.
* Receipt of any prescribed or over-the-counter (OTC) systemic, herbal (including St John's wort), or topical medication within 14 days of quizartinib administration, or any expectation of requiring use of such medication while participating in the study is prohibited.
* A positive drugs of abuse screen from a urine ethanol test (unless the drug is medically prescribed by a licensed health care provider) or alcohol breath test at Screening or at Check-in on Day -1 or a participant who will not agree to smoke ≤10 cigarettes or equivalent per day from Screening up to Enrollment, and is unable to be restricted to ≤5 cigarettes per day and for 6 hours post dose during their period of residence in the clinical unit
* Concomitant use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) and inhibitors of renal tubular secretion (eg, probenecid) within 14 days or 5 half-lives, if known, of the drugs, whichever is greater, prior to quizartinib administration
* Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome.
* Use of drugs with a risk of QT interval prolongation or torsade de pointes within 14 days of Day -1 (or 5 drug half-lives, if 5 drug half-lives are expected to exceed 14 days)
* Consumption of alcohol- and caffeine-containing beverages within 72 hours prior to check-in and during confinement
* Positive serology for hepatitis B surface antigen (HBsAg) and HCV (healthy subjects), hepatitis A virus (HAV) immunoglobulin M, or anti-human immunodeficiency virus (HIV) Type 1 and Type 2 (all participants)
* Current enrollment in or have not yet completed at least 30 days or 5 elimination half-lives, whichever is longer, since receiving an investigational device or product, or receipt of other investigational agents within 30 days of quizartinib

Additional Exclusion Criteria for Matched Healthy Participants:

* Any clinically relevant abnormality identified on the physical examination, ECG, vital signs, or laboratory tests at Screening
* Liver function (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase of liver origin, gamma-glutamyl transferase, and total bilirubin) test results above the upper limit of normal at Screening and during Enrollment on Day -2 are exclusionary. If transaminase levels are >2 × upper limit of normal (ULN) at Screening the participant will be excluded and cannot be rescreened

Additional Exclusion Criteria for Participants with Hepatic Impairment:

* Participants with active stage 3 or stage 4 encephalopathy
* Fluctuating or rapidly deteriorating hepatic function as indicated by recent history or worsening of clinical and/or laboratory signs of HI as judged by the investigator
* Participants with severe ascites and/or need of regular paracentesis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Advanced Pharma, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants who met all inclusion criteria and no exclusion criteria were enrolled from 22 Sep 2020 to 22 Jul 2021 at 3 clinics in the United States.
Pre-assignment Details: This study included a screening period up to 22 days prior to the enrolment and a 22 day in-clinic period, including screening.
Period: Overall Study
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (6.78) | 55.3 (3.88) | 56.2 (5.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration and was an observed value for the study.
Time Frame: Day 1 through 22: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 288, 360, 432, and 504 hours post-quizartinib dose
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng/mL | 86.2 (15.8) | 90.7 (17.7)
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; Statistical comparison was analyzed for Quizartinib; Test type: Other — Least squares (LS) means were calculated from an analysis of variance (ANOVA) model on log-transformed scale. The LS means for each treatment were back transformed from the log scale to provide estimates of the geometric means (GMS). The ratio (%) of GMS was calculated and 90% Confidence Intervals (CIs) for the ratio (%) of GMS were presented; Ratio (%) of Geometric LS Mean] = 95.1, 90% CI 2-sided [77.1 to 117] — For the comparison, the Moderate Hepatic Impairment treatment group represents the numerator and Normal Hepatic Function treatment group represents the denominator

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) for Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: Time of Maximum Plasma Concentration (Tmax) is defined as time of maximum observed plasma concentration and was an observed value from the study.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
hours | 4.0 [2.0 to 4.0] | 4.0 [2.0 to 4.0]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) for Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: Area Under the Plasma Concentration-Time Curve up to the Last Quantifiable Concentration Post-Dose (AUClast) is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method. Area Under the Plasma Concentration-Time Curve up to Infinity (AUCinf) is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity. AUClast and AUCinf was assessed.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng*h/mL
  AUClast | 7480 (2930) | 7720 (4750)
  AUCinf | 7880 (3540) | 8110 (5120)
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; AUClast statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean] = 109, 90% CI 2-sided [59.5 to 201] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; AUCinf statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean] = 109, 90% CI 2-sided [57.9 to 207] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Total Apparent Clearance (CL/F) for Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: Total Apparent Clearance (CL/F) is defined as total apparent clearance and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
L/h | 4.0 (1.9) | 5.0 (3.3)

5. Primary Outcome: Volume of Distribution in the Terminal Phase (Vz/F) for Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: Volume of Distribution in the Terminal Phase (Vz/F) is defined as volume of distribution in the terminal phase and was calculated using non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
Liters | 479 (121) | 577 (269)

6. Primary Outcome: Terminal Half-Life (t1/2) for Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: Terminal Elimination Half-Life (t1/2) is defined as terminal elimination half-life and was calculated using noncompartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
hours | 93.7 (36.0) | 96.3 (34.7)

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng/mL | 17.3 (12.1) | 24.7 (18.2)
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; Statistical comparison was analyzed for AC886; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 74.4, 90% CI 2-sided [32.0 to 173] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
hours | 7.00 [4.00 to 48.0] | 7.00 [4.00 to 72.0]

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) for Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set. For AUCinf, 1 participant was excluded from the Moderate Hepatic Impairment group where AUCinf based on extrapolation was greater than 20% and 1 participant was excluded from the Normal Hepatic Function group where Adjusted r-squared value was greater than 0.9.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng*h/mL
  AUClast | 2180 (1110) | 3240 (1280)
  AUCinf: number analyzed (Participants) | 5 | 5
  AUCinf | 2610 (878) | 3700 (1130)
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; AUClast statistical comparison was analyzed for AC886; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 62.5, 90% CI 2-sided [35.3 to 111] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; AUCinf statistical comparison was analyzed for AC886; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 69.9, 90% CI 2-sided [46.8 to 104] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Terminal Half-Life (t1/2) for Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 6
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
hours | 111.1 (48.7) | 81.4 (20.7)

11. Secondary Outcome: Metabolite to Parent Ratio (MPR) Based on Area Under the Curve for Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: AUCinf is defined as area under the plasma concentration-time curve from the time of dosing extrapolated to infinity and AUClast is defined as AUC from time 0 to the last measurable concentration, as calculated by the linear up-log down trapezoidal method. MPR is defined as a metabolite to parent ratio with metabolite as the numerator and the parent as the denominator. MPR corrected for molecular weight of AC886 of AUCinf and AUClast are reported and were calculated using non-compartmental analysis. AUClast and AUCinf was assessed.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ratio
  MPR AUClast | 0.363 (0.269) | 0.653 (0.496)
  MPR AUCinf: number analyzed (Participants) | 5 | 5
  MPR AUCinf | 0.428 (0.261) | 0.762 (0.467)

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Unbound Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng/mL | 0.412 (0.320) | 0.881 (0.692)
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; Statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 44.7, 90% CI 2-sided [18.0 to 111] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Unbound Quizartinib Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng*h/mL
  Unbound Quizartinib AUClast | 35.8 (30.4) | 84.5 (86.5)
  Unbound Quizartinib AUCinf | 37.4 (31.3) | 88.4 (90.0)
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; AUClast statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 51.5, 90% CI 2-sided [16.0 to 165] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants With Moderate Hepatic Impairment vs Control Participants With Normal Hepatic Function; AUCinf statistical comparison was analyzed for Quizartinib; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Mean = 51.5, 90% CI 2-sided [15.8 to 168] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Unbound Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set. Unbound AC886 concentration were below the level of quantification for 5 participants in the moderate hepatic impairment group and 2 participants in the normal hepatic function group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 1 | 4
ng/mL | 0.0553 (NA) — Not enough quantifiable data for estimation of standard deviation. | 0.0658 (0.0490)

15. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Unbound Active Metabolite AC886 Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter was assessed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
ng*h/mL
  Unbound AC886 AUClast | 4.06 (NA) — 5 participants had concentration below level of detection so there was not enough quantifiable data for estimation of standard deviation. | 7.17 (3.53)
  Unbound AC886 AUCinf: number analyzed (Participants) | 1 | 4
  Unbound AC886 AUCinf | 4.18 (NA) — Not enough quantifiable data for estimation of standard deviation. | 7.35 (3.56)

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Following Single Dose of Quizartinib in Participants With Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Description: A Treatment-Emergent Adverse Events (TEAE) is defined as any event not present prior to the initiation of the drug treatment of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment. Number of any TEAE that is related and unrelated to study medication is presented.
Time Frame: Baseline up to 30 days after last dose, up to 2 months
Population: TEAEs were assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of signing the informed consent form up to 30 days after last dose, up to 2 months.
Description: Adverse events were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within the 30 days after the last dose of the study drug.
Arm/Group | Participants With Moderate Hepatic Impairment | Control Participants With Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Moderate Hepatic Impairment (N=6) | Control Participants With Normal Hepatic Function (N=6)
Constipation (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04473664/Prot_SAP_000.pdf